CLINICAL TRIAL: NCT02138123
Title: Intraocular Lens-Shell Technique: An Adjustment of Surgical Procedure Makes Differences in Treating Dense Nucleus Cataract
Brief Title: Intraocular Lens-shell Technique in Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Ophthalmologist, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCPMOH2010-China5
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Cataract; Pseudoaphakia
Keywords: dense cataract; phacoemulsification; lens-shell technique; intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IOL-shell technique (Experimental): In this group, before the emulsification of the last nuclear fragment, cohesive viscoelastic material was injected below the nuclear fragment and a foldable IOL was implanted into the well inflated capsular bag posterior to the nuclear fragment. The remaining last piece of nuclear fragment was then emulsified and removed within the capsular bag.
  Interventions: Procedure: IOL-shell technique
- Conventional procedure (Active Comparator): In this group, a Sensar IOL (AMO Laboratories) was implanted in the capsular bag with the injector system after the lens material was completely removed. The nuclear fragmentation was performed using the Phaco-chop technique, which was then followed by ultrasound emulsification of the nuclear fragments piece by piece. Due to lack of cortical shell within the capsular bag, special care was taken to carry out the emulsification of the last nuclear fragment at a relatively more anterior anatomical position between the iris plan and the anterior chamber.
  Interventions: Procedure: Conventional procedure

INTERVENTIONS:
Procedure: IOL-shell technique — Phacoemulsification was performed with the same device and handpieces, using the same phaco chop technique as in the conventional procedure group. What was different was that before the emulsification of the last nuclear fragment, cohesive viscoelastic material was injected below the nuclear fragment and a foldable IOL was implanted into the well inflated capsular bag posterior to the nuclear fragment. The remaining last piece of nuclear fragment was then emulsified and removed within the capsular bag.
  Arms: IOL-shell technique
Procedure: Conventional procedure — In this procedure, a IOL was not implanted until all the nuclear fragments were removed.
  Arms: Conventional procedure

SUMMARY:
In this study, the investigators introduce a surgical procedure called "IOL-shell technique" in the purpose of reduce complications of surgeries for dense cataract, and report a prospective randomized controlled study aiming at assessing efficacy and safety of the IOL-shell technique, which showed that the new procedure offered a safer way for hard cataract surgery over the conventional phacoemulsification procedure without compromise in efficacy.

DETAILED DESCRIPTION:
A Prospective, randomized controlled study of 80 eyes with dense nucleus were enrolled. Patients were assigned to two groups: Group I: IOL was traditionally implanted after all nuclear fragments were completely removed, while in Group II, IOL was innovatively implanted in the bag before last residual nuclear fragment was removed. This novel adjusted surgical procedure, featured by using IOL as a protective barrier (named "IOL-shell technique"), not just as a refractive alternative, was conceptual different from the traditional step-by-step procedure. Clinical examinations including uncorrected visual acuity, central corneal thickness (CCT), temporal clear corneal thickness and the corneal endothelial cell density were carried out.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or above
* Dense cataract cases were defined as eyes in which the nuclear color was graded IV or V according to the Lens Opacities Classification System III (LOCS III). Special attention was paid in selecting cases without apparent posterior cortical layer.
* No central corneal opacification
* Pupil diameter >= 7 mm after full pharmacological dilation in preoperative assessment
* A preoperative central endothelial cell count of >= 1500 cells/mm2.

Exclusion Criteria:

* Participants with previous intraocular surgery
* Abnormal lens zonules
* Glaucoma
* High myopia (>-6.0 Diopters)
* Pseudoexfoliation
* Uveitis
* Diabetes mellitus
* Those who were not able to come for follow-up visits.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Central corneal endothelial cell loss | one month
  Central corneal endothelial cell loss was calculated by subtracting postoperative corneal endothelial cell density from the preoperative baseline level.

SECONDARY OUTCOMES:
central cornea thickness | one month
  The temporal corneal thickness and central corneal thickness were measured using the manual measurement scale in the scanning pictures of anterior segment optical coherence tomography preoperatively and at each postoperative visit.

OTHER OUTCOMES:
un-corrected visual acuity | one month
  The un-corrected visual acuity was measured and recorded using an Early Treatment Diabetic Retinopathy Study chart both before operation and at the 1st, 7th and 30th day after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center,Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Shah PA, Yoo S. Innovations in phacoemulsification technology. Curr Opin Ophthalmol. 2007 Feb;18(1):23-6. doi: 10.1097/ICU.0b013e328011f9d0. PMID 17159443
- [Background] Luo L, Lin H, He M, Congdon N, Yang Y, Liu Y. Clinical evaluation of three incision size-dependent phacoemulsification systems. Am J Ophthalmol. 2012 May;153(5):831-839.e2. doi: 10.1016/j.ajo.2011.10.034. Epub 2012 Feb 4. PMID 22310081
- [Background] Hwang HS, Kim EC, Kim MS. Drill-and-crack technique for nuclear disassembly of hard nucleus. J Cataract Refract Surg. 2010 Oct;36(10):1627-30. doi: 10.1016/j.jcrs.2010.08.003. PMID 20870105
- [Derived] Luo L, Lin H, Chen W, Qu B, Zhang X, Lin Z, Chen J, Liu Y. Intraocular lens-shell technique: adjustment of the surgical procedure leads to greater safety when treating dense nuclear cataracts. PLoS One. 2014 Nov 17;9(11):e112663. doi: 10.1371/journal.pone.0112663. eCollection 2014. PMID 25401512
- See also: Homepage of Zhongshan Ophthalmic Center — http://www.gzzoc.com/